CLINICAL TRIAL: NCT02402738
Title: Adjunctive Psychotherapy for Perinatal Bipolar Disorder
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: We chose to maximize this iterative treatment development study by terminating the pilot RCT in favor of enhancing an initial open trial (increased N 12 to 14)
Sponsor: Brown University (Other)
Collaborators: Butler Hospital (Other); Women and Infants Hospital of Rhode Island (Other); The Miriam Hospital (Other); Michigan State University (Other)
Responsible Party: Principal Investigator, Lauren M. Weinstock, PhD, Associate Professor (Research), Brown University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1R34MH102466-01A1 (NIH)
Record Dates: First submitted 2015-03-20; First posted 2015-03-30 (Estimated); Last update posted 2019-01-16 (Actual); Status verified 2019-01

CONDITIONS: Bipolar Disorder
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Interpersonal and Social Rhythm Therapy (Experimental): Participants may be randomized to receive up to 20 outpatient sessions of Interpersonal and Social Rhythm Therapy, provided as an adjunct to community treatment as usual. Intervention sessions begin during pregnancy and continue through 8 weeks postpartum.
  Interventions: Behavioral: Interpersonal and Social Rhythm Therapy
- Enhanced Treatment as Usual (Active Comparator): Those randomized to the Enhanced Treatment as Usual arm will follow their usual treatment plans in the community, with enhanced monitoring of symptoms and functioning through regular study assessments. With a release of information, we will provide community clinicians with a monthly standardized report that summarizes level of symptom severity and risk, designed to aid in continuity of care.
  Interventions: Behavioral: Enhanced Treatment as Usual

INTERVENTIONS:
Behavioral: Interpersonal and Social Rhythm Therapy
  Arms: Interpersonal and Social Rhythm Therapy
Behavioral: Enhanced Treatment as Usual
  Arms: Enhanced Treatment as Usual

SUMMARY:
Bipolar disorder (BD) is a serious, disabling, and highly recurrent illness. The perinatal period dramatically increases risk for mood episodes in women with BD, but pregnancy complicates pharmacologic treatment decisions and efficacy. This study will be the first to systematically develop and pilot test an adjunctive psychosocial intervention to assist in treatment of BD during the high-risk perinatal period.

DETAILED DESCRIPTION:
The perinatal period appears to be especially destabilizing for women with bipolar disorder (BD), with prospective studies revealing mood episode morbidity in up to 70% of pregnant women with the disorder, and risk of postpartum mania in as high as 50% of cases. There are clear negative sequelae of BD for mothers and their offspring, including gross maternal impairment, substantial risk for suicide, high risk of postpartum psychosis, and adverse childbirth outcomes. Yet data concerning the clinical management of BD during the perinatal period are strikingly limited. Pharmacotherapy is complicated due to known teratogenic risks of certain medications, the lack of safety data for others, and difficult treatment decisions, including the decision to discontinue pharmacotherapy, that women and clinicians face in light of limited data. Prophylactic mood stabilization has been widely recommended, yet data suggest that even among women with BD treated with medication, there remains significant risk of mood episode morbidity in the perinatal period. Given the pernicious course of BD in the perinatal period, adjunctive interventions aimed at improving clinical outcomes are critically needed. Interpersonal and Social Rhythm Therapy (IPSRT) is an adjunctive psychosocial intervention that may serve this need, as it: (a) incorporates key elements of Interpersonal Psychotherapy (IPT), which has a strong evidence base for treatment of perinatal depression in unipolar samples, (b) includes a behavioral intervention to stabilize the circadian rhythm disruption that may place perinatal women at high risk for mood and psychotic symptoms, (c) has established efficacy for the treatment of BD in non-perinatal samples, and (d) carries the promise of potential clinical benefit without additional fetal exposure. Yet there are no published studies evaluating the efficacy of IPSRT, or any psychosocial intervention, as an adjunct to pharmacotherapy for BD in the perinatal period. Given its many potential benefits, the primary aim of this R34 Exploratory Research Proposal (PAR-12-279) is to adapt and pilot IPSRT for perinatal women with BD. The development phase of this study will result in a treatment manual, training manual, and fidelity scales which will be tested in an open trial of 12 pregnant women with BD, treated through the early postpartum. The pilot phase will examine feasibility and acceptability of the proposed recruitment methods, research design, intervention, and interventionist training program by randomizing 40 pregnant women with BD to enhanced treatment as usual (E-TAU) or E-TAU + IPSRT, delivered through the early postpartum. Primary outcomes will be mood and psychotic symptoms up to 16 weeks postpartum. Additional outcomes include medication adherence, maternal functioning, and birth outcomes (secondary), and increased social support and circadian and social rhythm stability (tertiary). This pilot study will lay the groundwork for a larger, stage II clinical trial (R01) to evaluate the efficacy of this intervention for improving clinical and functional outcomes among this high risk, understudied population during the vulnerable transition from pregnancy to the postpartum period.

ELIGIBILITY:
Inclusion Criteria:

* DSM-5 diagnosis of bipolar I or bipolar II disorder
* at least moderately symptomatic (depression or manic symptoms) at time of study entry
* currently pregnant, up to 28 weeks gestation

Exclusion Criteria:

* presence of psychiatric symptoms severe enough to warrant inpatient hospitalization
* current psychotic symptoms
* active alcohol or substance use disorder
* cognitive deficits that preclude full understanding of study materials
* inability to understand English sufficiently well to understand consent or assessment instruments when read aloud
* plans to relocate within 8 months

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2014-04; Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Longitudinal Interval Follow-Up Evaluation (LIFE) | up to 16 weeks postpartum
  The LIFE is administered to calculate percent time symptomatic (with depression or mania symptoms) over the study period.
Quick Inventory of Depressive Symptomatology-Clinician Administered (QIDS-C) | up to 16 weeks postpartum
  The QIDS-C is administered to assess change in severity of depressive symptoms over study period.
Clinician-Administered Rating Scale for Mania (CARS-M) | up to 16 weeks postpartum
  The CARS-M is administered to assess change in severity of manic and psychotic symptoms over study period.

SECONDARY OUTCOMES:
Brief Quality of Life Scale for Bipolar Disorder (QoL.BD) | up to 16 weeks postpartum
Barkin Index of Maternal Functioning | up to 16 weeks postpartum
Medication Recommendation Tracking Form (MRTF) | up to 16 weeks postpartum

CONTACTS AND LOCATIONS:
Locations (1):
- Butler Hospital, Providence, Rhode Island, United States

REFERENCES:
- [Derived] Johansen SL, Robakis TK, Williams KE, Rasgon NL. Management of perinatal depression with non-drug interventions. BMJ. 2019 Feb 25;364:l322. doi: 10.1136/bmj.l322. PMID 30803997